CLINICAL TRIAL: NCT03496441
Title: The Relationship Between Intestinal Microbiota, Colorectal Cancer and Anastomotic Leakage After Colorectal Surgery: Pilot Study
Brief Title: Microbiota-anastomotic Leak Among Colorectal Surgery Patients : Pilot Study
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: CE 17.243
Record Dates: First submitted 2018-02-14; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Diseases; Microbiota; Anastomotic Leak
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For participants included in groups 1, 3 and 4, stool samples will be collected prior to surgery. For participants included in group 1 only, a stool sample will also be collected after surgery.
  For patients included in group 2, a sample of the digestive content (stool) will be collected during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Colorectal cancer patients who will undergo a surgical resection with digestive anastomosis. Fecal sample collection for analysis before and after surgery (2 samples).
  Interventions: Other: Fecal sample collection for analysis
- Group 2: Patients having undergone surgical resection with digestive anastomosis for colorectal cancer or inflammatory bowel disease, complicated by anastomotic leakage. Fecal sample collection for analysis after surgery, once the leak is confirmed.
  Interventions: Other: Fecal sample collection for analysis
- Group 3: Patients with uncomplicated hernia pathology, without gastrointestinal comorbidity to undergo a surgery to heal this hernia without involving a gastrointestinal resection. Fecal sample collection for analysis before surgery (1 sample).
  Interventions: Other: Fecal sample collection for analysis
- Group 4: Inflammatory bowel disease patients waiting for elective surgery involving gastrointestinal resection. Fecal sample collection for analysis during surgery, directly from the bowel content (1 sample).
  Interventions: Other: Fecal sample collection for analysis

INTERVENTIONS:
Other: Fecal sample collection for analysis — Fecal sample analysis will consist of the following procedure : Microbial DNA extraction, amplicon library construction, sequencing and analysis; Clustering MiSeq reads into operational taxonomic units (OTUs); Iron and heme measurements in the samples.

SUMMARY:
The study is based on the hypothesis that patients with postoperative anastomotic leakage have a different bacterial profile contributing to poor tissue healing, and that patients operated for colon cancer presumably have a different preoperative microbiota than healthy patients. This different composition is probably induced by the high heme level in the light intestinal tract that tumor spoliation generates.

The objective of the study is to evaluate the feasibility of a larger study to evaluate the difference between microbiota composition of patients with and without colorectal cancer, with inflammatory bowel disease and those with and without anastomotic leakage postoperatively of a colonic resection.

Stool samples will be taken from 20 patients, including 5 without intestinal pathology, 5 with colorectal cancer undergoing colorectal surgery, 5 with inflammatory bowel disease and 5 with anastomotic leakage after colectomy for colorectal cancer or inflammatory bowel disease.

The stool samples will be analyzed at CRCHUM to draw up a profile of the bacteria that make up the microbiota of each patient.

DETAILED DESCRIPTION:
No more details required.

ELIGIBILITY:
Inclusion Criteria:

ALL

* Informed consent obtained.
* Between 18 to 90 years old inclusive.
* Group 1 (colorectal cancer patients)

  * Patients with colorectal cancer confirmed with pathology results.
  * Oncological colon and / or rectal resection planned and performed by a surgeon from the digestive surgery department of the CHUM.
* Group 2 (anastomotic leak patients)

  * Patients with colorectal cancer confirmed with pathology and / or patients with inflammatory bowel disease.
  * Patients who underwent colonic and / or rectal surgical resection, complicated by an anastomotic leak in the postoperative period.
* Group 3 ("healthy" patients)

  * Patients with uncomplicated hernia pathology assessed externally in anticipation or after hernia repair surgery that does not involve gastrointestinal resection.
  * Patients with no history of colorectal neoplasia or surgical resection of the gastrointestinal tract.
* Group 4 (inflammatory bowel disease patients)

  * Patients with inflammatory bowel disease (IBD), waiting for elective surgery involving gastrointestinal resection.

Exclusion Criteria:

* Pregnancy.
* Class of the American Society of Anesthesiologists (ASA)> 3.
* Chemotherapy and / or pelvic and / or abdominal radiotherapy within 6 months prior to collection of the stool sample prior to surgery (group 3 with healthy patients only).
* Colonoscopy within 3 months prior to collection of the stool sample prior to surgery (group 3 with healthy patients only).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants included in groups 1,3 and 4 will be recruited at the outpatient clinic of the CHUM digestive surgery department, during the visit for evaluation prior surgery.
  Participants included in group 2 will be recruited during the post surgery period, during their hospitalization in the department of digestive surgery of the CHUM.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of patients' recruitment | 3 months
  Evaluate if we can recruit all required patients easily ; 20 patients total and 5 patients per group (Yes or No).
Evaluate the feasibility of fecal samples' analysis | 3 months
  Evaluate if we can easily perform the fecal sample analysis with the establish procedures (Yes or No).

SECONDARY OUTCOMES:
Evaluation the presence of a correlation between fecal microbiota composition and the risk of anastomotic leak. | 6 months
  If it is possible to obtain results from the fecal samples' analysis, a possible correlation in the results will be evaluate.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Richard, MD, FRCSC, Principal Investigator — Centre Hospitalier Universitaire de Montreal
Locations (1):
- Centre Hospitalier Universitaire de Montreal (CHUM), Montreal, Quebec, Canada